CLINICAL TRIAL: NCT03023098
Title: Drug-eluting Balloon vs. Conventional Balloon in the Treatment of (re)Stenosis - a Randomized Prospective Study
Acronym: DRECOREST1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Maarit Venermo, Professor of Vascular Surgery, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DRECOREST1 - Jan 23rd 2013
Record Dates: First submitted 2017-01-12; First posted 2017-01-18 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Peripheral Artery Occlusive Disease; Peripheral Artery Restenosis; Peripheral Artery Stenosis
Keywords: Restenosis; Drug-eluting balloon; Vein graft
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1 | interventions — Angioplasty; Angioplasty, Balloon

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug-eluting balloon (Experimental)
  Interventions: Device: Drug-eluting balloon
- Conventional PTA (Active Comparator)
  Interventions: Device: Conventional PTA

INTERVENTIONS:
Device: Conventional PTA — After passing the stenosis it is dilated with a conventional balloon. The patient is randomized to a second dilatation with a conventional balloon
  Other Names: PTA (percutaneous transluminal angioplasty); Balloon angioplasty
  Arms: Conventional PTA
Device: Drug-eluting balloon — After passing the stenosis it is dilated with a conventional balloon. The patient is randomized to a second dilatation with a drug-eluting balloon
  Other Names: DEB
  Arms: Drug-eluting balloon

SUMMARY:
The purpose of this study is to determine whether the use of drug-eluting balloons is effective in the treatment of (re)stenosis in bypass vein grafts.

DETAILED DESCRIPTION:
Drug-eluting devices have proved beneficial in the treatment of stenosis in native coronary and lower limb arteries. Stenosis and restenosis is a known problem in bypass vein grafts, and drug-eluting devices might be beneficial in this field as well.

In the procedure a conventional balloon is passed through the stenosis which is then dilated. After this patients are randomized before a second dilatation with either a conventional balloon or a drug-coated balloon.

The stenosis is evaluated preoperatively and followed up by means of ultrasound by a vascular technician. Follow-up will end at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Any venous bypass with stenosis warranting intervention

Exclusion Criteria:

* Previous PTA with drug-eluting balloon, thrombolysis, coagulopathy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-01; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
TLR (Target lesion revascularization) | 12 months
  Any reintervention to the same lesion.
Graft occlusion | 0-12 months
  Occlusion of the bypass graft

SECONDARY OUTCOMES:
Major amputation | 0-12 months
  Above or below knee amputation of the treated leg
Death | 0-12 months

OTHER OUTCOMES:
Primary assisted patency | 0-12 months
  Patency of the graft after TLR

CONTACTS AND LOCATIONS:
Overall Officials: Maarit Venermo, M.D., Ph.D., Study Director — Helsinki University Hospital, Dept. of Vascular Surgery
Locations (1):
- Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bjorkman P, Kokkonen T, Alback A, Venermo M. Drug-Coated versus Plain Balloon Angioplasty in Bypass Vein Grafts (the DRECOREST I-Study). Ann Vasc Surg. 2019 Feb;55:36-44. doi: 10.1016/j.avsg.2018.04.042. Epub 2018 Aug 6. PMID 30092443